CLINICAL TRIAL: NCT02289014
Title: Web-based Stress Management for Newly Diagnosed Cancer Patients (STREAM-1): A Randomized, Wait-list Controlled Intervention Study
Brief Title: Web-based Stress Management for Newly Diagnosed Cancer Patients (STREAM-1)
Acronym: STREAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Krebsforschung Schweiz, Bern, Switzerland (Other); Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KFS-3260-08-2013
Record Dates: First submitted 2014-10-09; First posted 2014-11-13 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Psychological Distress; Cancer
Keywords: online intervention; stress management; cognitive behavioral therapy; acceptance and mindfulness based intervention
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wait-list control group (No Intervention): Wait-list control group
- Active treatment group (Experimental): online stress Management program
  Interventions: Other: online stress Management program

INTERVENTIONS:
Other: online stress Management program — Active treatment group
  Arms: Active treatment group

SUMMARY:
Many cancer patients experience their illness as substantial psychological burden. About half of the cancer patients suffer from severe stress symptoms and around one third of the patients fulfill the criteria for a clinically relevant psychological disorder (mainly anxiety disorder and/or major depression). Studies show, that a high level of distress in cancer patients is associated with more side effects of and a reduced compliance for oncological treatment.

Today, the efficacy of psycho-oncological interventions is well studied and proven. Besides the reduction of levels of anxiety, distress and depression, psycho-oncological support facilitates dealing with physical complaints and increases quality of life. Yet, psycho-oncological support is rarely utilized by male patients and insufficiently accessible for many patients (i.a. lack of supply in the respective area, cost issues).

The internet overcomes some of these barriers, as it can be used independently of time and location. Internet-based therapies are therefore a growing field of interest in research and there is evidence for treatment efficacy for several psychological disorders. Moreover effect sizes of traditional face-to-face and interactive web-based interventions are comparable. However, web-based interventions for cancer patients are still scarce. The present research project therefore develops a comprehensive stress management program accessible for a vast number of cancer patients. The study targets primarily to evaluate the feasibility of the program (technical, organizational feasibility, accessibility). In addition, the preliminary efficacy of the program will be analyzed in order to adapt future programs for specific patient groups.

DETAILED DESCRIPTION:
The present study is designed as a randomized controlled wait-list intervention study. Within 12 weeks of the start of anti-cancer treatment, patients will be randomly assigned to the web-based stress management intervention or a wait-list control condition.

Inclusion criteria:

Patients with any kind of newly diagnosed cancer undergoing first Treatment regardless of the Setting. Patients undergoing first treatment for newly diagnosed relapse of cancer, who have received prior curatively-intended Treatment.

Inclusion is allowed immediately prior to or within 12 weeks of the start of treatment. If surgery was performed initially and is followed by systemic treatment or radiotherapy, start of systemic treatment or radiotherapy is counted as first treatment. Prior treatment -including chemotherapy- for a different, prior malignant tumor is allowed. Concomitant participation in an experimental therapeutic drug trial is allowed. Age >18 years. Command of the German language. Internet access and basic computer skills. Life expectancy of >6 months.

Exclusion criteria:

Patients undergoing second- or further line treatment. Patients treated with surgery only. Patients participating in a concomitant psychological intervention trial

ELIGIBILITY:
Inclusion Criteria:

* Patients with any kind of newly diagnosed cancer undergoing first treatment (including radiotherapy, hormonal treatment, targeted therapies, chemotherapy or combined-modality treatment) regardless of the setting (adjuvant treatment, curative treatment, palliative first-line treatment)
* Patients with newly diagnosed relapse of cancer, who had received prior curatively-intended treatment
* Inclusion is allowed immediately prior to or within 12 weeks of the start of treatment
* Patients must have cytologically or histologically proven diagnosis of malignant disease (either at diagnosis or at relapse)
* Prior treatment -including chemotherapy- for a different, prior malignant tumor is allowed
* Concomitant participation in an experimental therapeutic drug trial is allowed
* Age >18 years
* Command of the German language
* Internet access and basic computer skills
* Life expectancy of >6 months

Exclusion Criteria:

* Patients undergoing palliative second- or further line chemotherapy treatment
* Patients treated with surgery only
* Patients participating in a concomitant psychological intervention trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2014-01; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Dropout rate during the internet-based recruitment procedure | Measures assessed at time point of recruitment
Characteristics (Sociodemographic and medical history; i.e. age, gender, education, cancer diagnosis and cancer treatment) of the population willing to participate in an online stress management program shortly after diagnosis of cancer | Measures assessed at time point of recruitment
Number of participants who completed at least 6 out of 8 modules, i.e. 75 % of each module | participants will be followed for the duration of the intervention, an expected average of 8 weeks
Working Alliance scores on the Working Alliance (WAI) Questionnaire | participants will be followed for the duration of the intervention, an expected average of 8 weeks
Usability scores on the System Usability Scale (SUS) | participants will be followed for the duration of the intervention, an expected average of 8 weeks
Client satisfaction on the Client Satisfaction Questionnaire-8 (CSQ-8) | Measures assessed after 8 weeks
  German Version of the Client Satisfaction Questionnaire: Fragebogen zur Messung der Patientenzufriedenheit (ZUF-8) will be used

SECONDARY OUTCOMES:
Psychological distress on the Distress Thermometer (visual analogue scale) | Change measures (e.g., "baseline, 8 weeks")
Anxiety and Depression scores on the Hospital Anxiety and Depression Scale (HADS) | Change measures (e.g., "baseline, 8 weeks")
Quality of life and fatigue scores on the Functional Assessment in Cancer Therapy-Fatigue (FACT-F) | hange measures (e.g., "baseline, 8 weeks")
Avoidance and psychological inflexibility scores on the Acceptance and Action questionnaire (AAQ) | ange measures (e.g., "baseline, 8 weeks")
  German Version of the Acceptance and Action questionnaire: Fragebogen zur Akzeptanz und Handeln (FAH II) will be used

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Urech, Dr. phil., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Urech C, Grossert A, Alder J, Scherer S, Handschin B, Kasenda B, Borislavova B, Degen S, Erb J, Faessler A, Gattlen L, Schibli S, Werndli C, Gaab J, Berger T, Zumbrunn T, Hess V. Web-Based Stress Management for Newly Diagnosed Patients With Cancer (STREAM): A Randomized, Wait-List Controlled Intervention Study. J Clin Oncol. 2018 Mar 10;36(8):780-788. doi: 10.1200/JCO.2017.74.8491. Epub 2018 Jan 25. PMID 29369731
- [Derived] Grossert A, Urech C, Alder J, Gaab J, Berger T, Hess V. Web-based stress management for newly diagnosed cancer patients (STREAM-1): a randomized, wait-list controlled intervention study. BMC Cancer. 2016 Nov 3;16(1):838. doi: 10.1186/s12885-016-2866-0. PMID 27809796